CLINICAL TRIAL: NCT06793150
Title: Comparison of the Effects of Opioid-Based Anesthesia Versus Opioid-Free Anesthesia on Postoperative Cognitive Dysfunction in Transsphenoidal Pituitary Surgeries
Brief Title: Postoperative Cognitive Dysfunction in Transsphenoidal Pituitary Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Gökçe Çile Özer, principal investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-AR-GÇÖ-01
Record Dates: First submitted 2024-07-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Dysfunction; Opioid Free Anesthesia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Remifentanil; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: group d maintaiance with dexmedetomidine group r maintainence with remifentanile
Who Masked: Participant
Masking Description: group d maintaiance with dexmedetomidine group r maintainence with remifentanile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group d (Active Comparator): group d anesthesia maintaiance with dexmedetomidine
  Interventions: Drug: dexmedetomidin
- group r (Active Comparator): group r anesthesia maintainence with remifentanile
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — A comparison will be made by maintaining one group with remifentanil and the other with dexmedetomidine.
  Other Names: ultiva
  Arms: group r
Drug: dexmedetomidin — A comparison will be made by maintaining one group with remifentanil and the other with dexmedetomidine.
  Other Names: sedadomid
  Arms: group d

SUMMARY:
In this study, the patients undergoing pituitary surgery in our clinic have examined in two groups. In the first group, anesthesia maintenance was provided with remifentanil and propofol infusion. In the second group, anesthesia maintenance was provided with dexmedetomidine and propofol infusion. Demographic data, vital signs during the operation, wake-up time, extubation time, and drug consumption amounts were recorded. The mini-mental test was applied preoperatively, 24 hours postoperatively, and 3 weeks postoperatively to examine whether there is a difference in cognitive dysfunction between the two groups.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction refers to disorders affecting orientation, attention, perception, consciousness, and judgment that develop after surgery. It is a common postoperative complication and a serious threat to the quality of life, particularly for elderly patients. Strategies to prevent surgery and anesthesia-induced cognitive dysfunction are being investigated, considering the choice and depth of anesthesia, perioperative anesthetic and other drugs, and surgical strategy.

Opioid-free anesthesia involves the administration of intraoperative anesthesia without the use of intraoperative opioids. Currently available non-opioid drugs include acetaminophen, nonsteroidal anti-inflammatory drugs (NSAIDs) (ketorolac, ibuprofen, celecoxib), alpha-2 agonists (dexmedetomidine, clonidine, tizanidine), and N-methyl-D-aspartate (NMDA) receptor antagonists (ketamine). Dexmedetomidine (DEX) is an alpha-2 adrenoceptor agonist with a selectivity ratio of 1600:1 (α2:α1). It promotes sedation by acting on the α2 receptors of the locus coeruleus and produces analgesia by reducing the release of substance P in the spinal cord dorsal horn.

The goals of opioid use during anesthesia are to reduce the need for hypnotic agents and provide effective analgesia. However, the potential side effects of opioids can be described as having a threefold negative impact, ranging from sudden adverse reactions in the patient to the long-term sequelae of chronic effects.

In this study, the patients undergoing pituitary surgery in our clinic have examined in two groups. In the first group, anesthesia maintenance was provided with remifentanil and propofol infusion. In the second group, anesthesia maintenance was provided with dexmedetomidine and propofol infusion. Demographic data, vital signs during the operation, wake-up time, extubation time, and drug consumption amounts were recorded. The mini-mental test was applied preoperatively, 24 hours postoperatively, and 3 weeks postoperatively to examine whether there is a difference in cognitive dysfunction between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transsphenoidal pituitary elective surgery
* Patients classified as ASA (American Society of Anesthesiologists) physical status classification I-III
* Patients aged between 18 and 65 years

Exclusion Criteria:

* Patients scheduled for emergency surgery
* Patients classified as ASA (American Society of Anesthesiologists) physical status classification IV-V
* Patients with psychiatric disorders
* Patients with a history of stroke, dementia, electrolyte disturbances, or serious liver and/or kidney disease
* Patients with a history of substance abuse"

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
cognitive dysfunction | preoperative, postoperative 24th hour and 3rd week
  Our primary objective is comparing postoperative cognitive dysfunction using the Mini-Mental State Examination after anesthesia 24 hours and 3 weeks after surgery

SECONDARY OUTCOMES:
comparing anesthesia and opioid free anesthesia | preoperative, postoperative 24th hour and 3rd week
  Our secondary objective is to compare the times of eye opening and extubation after opioid free anesthesia and anesthesia with opioid.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin X, Chen Y, Zhang P, Chen G, Zhou Y, Yu X. The potential mechanism of postoperative cognitive dysfunction in older people. Exp Gerontol. 2020 Feb;130:110791. doi: 10.1016/j.exger.2019.110791. Epub 2019 Nov 23. PMID 31765741
- [Background] Kotekar N, Shenkar A, Nagaraj R. Postoperative cognitive dysfunction - current preventive strategies. Clin Interv Aging. 2018 Nov 8;13:2267-2273. doi: 10.2147/CIA.S133896. eCollection 2018. PMID 30519008
- [Background] Chia PA, Cannesson M, Bui CCM. Opioid free anesthesia: feasible? Curr Opin Anaesthesiol. 2020 Aug;33(4):512-517. doi: 10.1097/ACO.0000000000000878. PMID 32530891